CLINICAL TRIAL: NCT06278064
Title: Plasma Extracellular Vesicle Quantitative Proteomic Analysis for Early Diagnosis of Upper Gastrointestinal Cancers
Brief Title: Exosome-based Liquid Biopsies for Upper Gastrointestinal Cancers Diagnosis
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Min Li, Deputy Director of Science and Technology Department, Beijing Friendship Hospital
Other Study IDs: BFHHZML20240006
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer; Esophagus Cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Only proteins will be detected and analyzed in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Gastric cancer group: Patients diagnosed with gastric cancer, including early gastric cancer and advanced gastric cancer
  Interventions: Other: Gastric Cancer
- esophagus cancer group: Patients diagnosed with esophagus cancer, including early esophagus cancer and advanced esophagus cancer
  Interventions: Other: Esophagus Cancer
- Non-cancer group: Patients diagnosed with benign upper gastrointestinal diseases or healthy controls

INTERVENTIONS:
Other: Gastric Cancer — Patients diagnosed with gastric cancer, including early stage gastric and advanced gastric cancer
  Groups: Gastric cancer group
Other: Esophagus Cancer — Patients diagnosed with esophagus cancer, including early esophagus gastric and advanced esophagus cancer
  Groups: esophagus cancer group

SUMMARY:
This study constitutes a case-control investigation employing a retrospective approach. Plasma samples from individuals with esophageal cancer, benign esophageal diseases, gastric cancer, benign gastric diseases, and a healthy control group were systematically collected. Advanced Data-Independent Acquisition (DIA) proteomics and single-vesicle membrane protein detection techniques were employed to quantify protein content within exosomes. Specific protein biomarkers indicative of early-stage upper gastrointestinal tumors were identified. External validation of these protein markers was conducted using Parallel Reaction Monitoring (PRM) technology on an independent validation cohort. The objective is to establish protein marker predictions for early diagnosis of upper gastrointestinal tumors and prognostication of therapeutic efficacy.

DETAILED DESCRIPTION:
This study employs a multicenter, retrospective cohort design, collecting and analyzing plasma and tissue exosome protein data from patients with upper gastrointestinal tumors (Stage I-II), upper gastrointestinal benign diseases, and a healthy control group who have visited Beijing Friendship Hospital, and other relevant sub-center hospitals over the past five years. Concurrently, relevant clinical and pathological information is recorded.

Samples from the training cohort undergo traditional quantitative exosome proteomic analysis (Data-Independent Acquisition, DIA) and single-vesicle membrane protein analysis (PBA). A comprehensive upper gastrointestinal tumor-specific exosome protein database is constructed, incorporating extensive information. Subsequently, bioinformatics methods are employed to conduct in-depth analysis of the extensive protein data, screening for proteins with high specificity for upper gastrointestinal tumors, capable of direct detection on the exosome membrane surface. By establishing and evaluating diagnostic models, we aim to quantify the diagnostic potential of these markers, providing a scientific basis for future early screening methods for upper gastrointestinal tumors.

Finally, external validation of these protein markers in an independent validation cohort ensures their reliability and stability across different patient populations. The academic significance of this research lies in its thorough exploration of exosome proteomics in early cancer diagnosis, offering potential innovative breakthroughs for academic progress and clinical practice in this field.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of upper gastrointestinal cancers or benign upper gastrointestinal diseases through gastroscopy and pathological examination.
* Collection of plasma samples prior to surgical treatment.
* Availability of complete clinical data.

Exclusion Criteria:

* Previous reception of anti-tumor treatments (including radiotherapy, chemotherapy, etc.) before blood collection.
* Coexistence of other systemic tumors.
* Absence of plasma sample collection before surgical treatment.
* Incomplete clinical data.
* Pregnancy status

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population included a range of subjects with upper gastrointestinal cancers and diseases, including patients with malignant and benign upper gastrointestinal diseases and healthy controls, who were admitted to the main study center and other collaborating sub-center hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 562 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Plasma proteins in patients with gastric cancer | Before receiving treatment for gastric cancer
  The outcome will be tested by Data-Independent Acquisition (DIA) proteomics technology
Plasma proteins in patients with esophagus cancer | Before receiving treatment for esophagus cancer
  The outcome will be tested by Data-Independent Acquisition (DIA) proteomics technology

CONTACTS AND LOCATIONS:
Overall Officials: Li Min, Ph.D., Principal Investigator — Beijing Friendship Hospital
Locations (3):
- China (3):
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing